CLINICAL TRIAL: NCT02395107
Title: Left Atrial Volume Index - Impact on LV Remodeling, LV Function and Functional Capacity in Asymptomatic Aortic Valve Stenosis
Brief Title: Left Atrial Volume Index in Asymptomatic Aortic Stenosis
Acronym: LAVIAS
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Nicolaj Lyhne Christensen, MD, Odense University Hospital
Other Study IDs: S-20130067
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Aortic Valve Stenosis; Heart Failure
Keywords: Aortic Valve Stenosis; Functional Capacity; Cardiomyopathies; Endomyocardial Fibrosis; Cardiovascular Diseases; Heart Diseases; Heart Valve Diseases; Atrial Fibrillation; Hypertrophy; Hypertrophy, Left Ventricular; Diastology
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure; Cardiomyopathies; Endomyocardial Fibrosis; Cardiovascular Diseases; Heart Diseases; Heart Valve Diseases; Atrial Fibrillation; Hypertrophy; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Aortic stenosis results in increased filling pressures of the heart. Size and function of the left atrium may be a marker for more advanced heart disease (heart failure) in patients with severe aortic stenosis, not presenting any apparent symptoms.

The goal of this study is to establish the importance and possible implications of left atrial dilation in asymptomatic patients with aortic valve stenosis.

DETAILED DESCRIPTION:
Aortic valve stenosis (AS) is the most common valvular disease in the western world. Mild and moderate AS generally is well tolerated severe AS is associated with considerable morbidity and mortality.

The consequence of AS is increased pressure load on the left ventricle, which causes changes in the ventricular function and structure (Left ventricular remodeling, hypertrophy, fibrosis).

With longstanding elevated filling pressures the left atrium will dilate and heart failure symptoms will develop.

When apparent, symptoms of heart failure, in AS are associated with high mortality rate and aortic valve replacement (AVR) is recommended.

The clinical assessment of heart failure symptoms in AS is however challenging particularly in the elderly, as symptoms progress slowly and may mimic age related fragility.

In this observational study, the goal is to investigate the importance and possible implications of left atrial dilation and heart failure among 100 patients with asymptomatic severe aortic stenosis. Participants undergo echocardiographic evaluation for diastolic heart failure and we assess myocardial fibrosis using magnetic resonance imaging and exercise testing with invasive hemodynamic monitoring (right heart catheterization).

LA dilatation may potentially identify patients likely benefiting of early surgery. The importance and possible implications of LA dilatation in asymptomatic AS patients has however not yet been established.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic severe aortic stenosis (Vmax > 3.5 m/sec and aortic valve area < 1 cm2).

Exclusion Criteria:

* Moderate LV systolic dysfunction (LVEF < 50%)
* Concomitant moderate-severe aortic valve regurgitation
* Concomitant moderate-severe mitral valve regurgitation
* Moderate to severe nephropathy
* Chronic or persistent atrial fibrillation
* Implanted pacemaker or cardio defibrillator
* Disability to exercise testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe asymptomatic aortic stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 2 years
  Differences in functional capacity reflected by atrial size. An incremental maximal exersice test to determine maximal whole-body oxygen uptake (VO2-max) will be performed. On a cycle ergometer VO2 and VCO2 are measured continuously with a breath-by-breath pulmonary exchange system. Following the warm up, the resistance is increased every 2 minutes for 3 bouts, where after the resistance increases every minute (10% increments in VO2-max). The test is terminated 30 seconds after the subjects are unable to maintain 60 revolutions pr. min, but are still able to bike. A horizontal plateau on the oxygen uptake graph demarks the maximal oxygen uptake in liters pr. min. This is divided by their body mass, to obtain maximal oxygen uptake pr. mass unit pr. time unit.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob E Møller, MD PhD DMsc, Study Director — Odense University Hospital; Jordi S Dahl, MD PhD, Study Chair — Odense University Hospital; Lars M Videbæk, MD PhD, Study Chair — Odense University Hospital; Eva Søndergaard, MD PhD, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Derived] Andersen MJ, Wolsk E, Bakkestrom R, Christensen N, Carter-Storch R, Omar M, Dahl JS, Frederiksen PH, Borlaug B, Gustafsson F, Hassager C, Moller JE. Pressure-flow responses to exercise in aortic stenosis, mitral regurgitation and diastolic dysfunction. Heart. 2022 Nov 10;108(23):1895-1903. doi: 10.1136/heartjnl-2022-321204. PMID 36356959
- [Derived] Carter-Storch R, Mortensen NSB, Christensen NL, Ali M, Laursen KB, Pellikka PA, Moller JE, Dahl JS. First-phase ejection fraction: association with remodelling and outcome in aortic valve stenosis. Open Heart. 2021 Feb;8(1):e001543. doi: 10.1136/openhrt-2020-001543. PMID 33574022
- [Derived] Christensen NL, Dahl JS, Carter-Storch R, Bakkestrom R, Jensen K, Steffensen FH, Sondergaard EV, Videbaek L, Moller JE. Association Between Left Atrial Dilatation and Invasive Hemodynamics at Rest and During Exercise in Asymptomatic Aortic Stenosis. Circ Cardiovasc Imaging. 2016 Oct;9(10):e005156. doi: 10.1161/CIRCIMAGING.116.005156. PMID 27894069